CLINICAL TRIAL: NCT00005197
Title: Predictors of Perioperative Cardiac Morbidity
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1076; R01HL036744 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Myocardial Infarction; Ventricular Arrhythmia; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Myocardial Infarction; Coronary Disease

SUMMARY:
To determine the predictors of perioperative cardiac morbidity and mortality in patients at high risk who underwent major noncardiac surgery with general anesthesia.

DETAILED DESCRIPTION:
BACKGROUND:

Of the 25 million patients who undergo noncardiac surgery in the United States each year, approximately three million have or are at risk of having coronary artery disease. Despite advances in the diagnosis and therapy of coronary artery disease, approximately 50,000 of these patients have a perioperative myocardial infarction, and more than half of the 40,000 deaths after surgery are caused by cardiac events. For perioperative myocardial infarction alone, health care costs exceeded $500 million per year in the 1980s. Determining the risk factors for adverse postoperative cardiac outcomes allowed the development of preventive strategies and the efficient allocation of health care resources.

DESIGN NARRATIVE:

Historical, clinical, laboratory, and physiologic data on the subjects were collected during hospitalization for major elective noncardiac surgery with general anesthesia and for six to 24 months after surgery. Myocardial ischemia was assessed by continuous electrocardiographic monitoring, beginning two days before surgery and continuing for two days after. The study published many findings under the title Study of Perioperative Ischemia.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-12; Study Completion 1991-11 (Actual)

REFERENCES:
- [Background] Mangano DT, Browner WS, Hollenberg M, London MJ, Tubau JF, Tateo IM. Association of perioperative myocardial ischemia with cardiac morbidity and mortality in men undergoing noncardiac surgery. The Study of Perioperative Ischemia Research Group. N Engl J Med. 1990 Dec 27;323(26):1781-8. doi: 10.1056/NEJM199012273232601. PMID 2247116
- [Background] Mangano DT, Hollenberg M, Fegert G, Meyer ML, London MJ, Tubau JF, Krupski WC. Perioperative myocardial ischemia in patients undergoing noncardiac surgery--I: Incidence and severity during the 4 day perioperative period. The Study of Perioperative Ischemia (SPI) Research Group. J Am Coll Cardiol. 1991 Mar 15;17(4):843-50. doi: 10.1016/0735-1097(91)90863-5. PMID 1999618
- [Background] Mangano DT, Wong MG, London MJ, Tubau JF, Rapp JA. Perioperative myocardial ischemia in patients undergoing noncardiac surgery--II: Incidence and severity during the 1st week after surgery. The Study of Perioperative Ischemia (SPI) Research Group. J Am Coll Cardiol. 1991 Mar 15;17(4):851-7. doi: 10.1016/0735-1097(91)90864-6. PMID 1999619
- [Background] Smith RC, Leung JM, Keith FM, Merrick S, Mangano DT. Ventricular dysrhythmias in patients undergoing coronary artery bypass graft surgery: incidence, characteristics, and prognostic importance. Study of Perioperative Ischemia (SPI) Research Group. Am Heart J. 1992 Jan;123(1):73-81. doi: 10.1016/0002-8703(92)90749-l. PMID 1370363
- [Background] Mangano DT, Siliciano D, Hollenberg M, Leung JM, Browner WS, Goehner P, Merrick S, Verrier E. Postoperative myocardial ischemia. Therapeutic trials using intensive analgesia following surgery. The Study of Perioperative Ischemia (SPI) Research Group. Anesthesiology. 1992 Mar;76(3):342-53. PMID 1531742
- [Background] Browner WS, Li J, Mangano DT. In-hospital and long-term mortality in male veterans following noncardiac surgery. The Study of Perioperative Ischemia Research Group. JAMA. 1992 Jul 8;268(2):228-32. PMID 1608142
- [Background] O'Kelly B, Browner WS, Massie B, Tubau J, Ngo L, Mangano DT. Ventricular arrhythmias in patients undergoing noncardiac surgery. The Study of Perioperative Ischemia Research Group. JAMA. 1992 Jul 8;268(2):217-21. doi: 10.1001/jama.268.2.217. PMID 1608140
- [Background] Krupski WC, Layug EL, Reilly LM, Rapp JH, Mangano DT. Comparison of cardiac morbidity between aortic and infrainguinal operations. Study of Perioperative Ischemia (SPI) Research Group. J Vasc Surg. 1992 Feb;15(2):354-63; discussion 364-5. PMID 1735896
- [Background] Mangano DT, London MJ, Tubau JF, Browner WS, Hollenberg M, Krupski W, Layug EL, Massie B. Dipyridamole thallium-201 scintigraphy as a preoperative screening test. A reexamination of its predictive potential. Study of Perioperative Ischemia Research Group. Circulation. 1991 Aug;84(2):493-502. doi: 10.1161/01.cir.84.2.493. PMID 1860194
- [Background] Mangano DT. Myocardial ischemia following surgery: preliminary findings. Study of Perioperative Ischemia (SPI) Research Group. J Card Surg. 1990 Sep;5(3 Suppl):288-93. doi: 10.1111/jocs.1990.5.3s.288. PMID 2133859
- [Background] Mangano DT. Dynamic predictors of perioperative risk. Study of Perioperative Ischemia (SPI) Research Group. J Card Surg. 1990 Sep;5(3 Suppl):231-6. doi: 10.1111/jocs.1990.5.3s.231. PMID 2133848
- [Background] Leung JM, Hollenberg M, O'Kelly BF, Kao A, Mangano DT. Effects of steal-prone anatomy on intraoperative myocardial ischemia. The SPI Research Group. J Am Coll Cardiol. 1992 Nov 1;20(5):1205-12. doi: 10.1016/0735-1097(92)90379-2. PMID 1401623
- [Background] Hollenberg M, Mangano DT, Browner WS, London MJ, Tubau JF, Tateo IM. Predictors of postoperative myocardial ischemia in patients undergoing noncardiac surgery. The Study of Perioperative Ischemia Research Group. JAMA. 1992 Jul 8;268(2):205-9. PMID 1535109
- [Background] Simon JA, Browner WS, Mangano DT. Predictors of smoking relapse after noncardiac surgery. Study of Perioperative Ischemia (SPI) Research Group. Am J Public Health. 1992 Sep;82(9):1235-7. doi: 10.2105/ajph.82.9.1235. PMID 1503164
- [Background] Mangano DT, Browner WS, Hollenberg M, Li J, Tateo IM. Long-term cardiac prognosis following noncardiac surgery. The Study of Perioperative Ischemia Research Group. JAMA. 1992 Jul 8;268(2):233-9. doi: 10.1001/jama.268.2.233. PMID 1608143
- [Background] Eisenberg MJ, London MJ, Leung JM, Browner WS, Hollenberg M, Tubau JF, Tateo IM, Schiller NB, Mangano DT. Monitoring for myocardial ischemia during noncardiac surgery. A technology assessment of transesophageal echocardiography and 12-lead electrocardiography. The Study of Perioperative Ischemia Research Group. JAMA. 1992 Jul 8;268(2):210-6. doi: 10.1001/jama.268.2.210. PMID 1608139
- [Background] Leung JM, Goehner P, O'Kelly BF, Hollenberg M, Pineda N, Cason BA, Mangano DT. Isoflurane anesthesia and myocardial ischemia: comparative risk versus sufentanil anesthesia in patients undergoing coronary artery bypass graft surgery. The SPI (Study of Perioperative Ischemia) Research Group. Anesthesiology. 1991 May;74(5):838-47. PMID 1826989
- [Background] Smith RC, Leung JM, Mangano DT. Postoperative myocardial ischemia in patients undergoing coronary artery bypass graft surgery. S.P.I. Research Group. Anesthesiology. 1991 Mar;74(3):464-73. doi: 10.1097/00000542-199103000-00013. PMID 2001026
- [Background] Leung JM, O'Kelly BF, Mangano DT. Relationship of regional wall motion abnormalities to hemodynamic indices of myocardial oxygen supply and demand in patients undergoing CABG surgery. Anesthesiology. 1990 Nov;73(5):802-14. doi: 10.1097/00000542-199011000-00002. PMID 2240670
- [Background] London MJ, Tubau JF, Wong MG, Layug E, Hollenberg M, Krupski WC, Rapp JH, Browner WS, Mangano DT. The "natural history" of segmental wall motion abnormalities in patients undergoing noncardiac surgery. S.P.I. Research Group. Anesthesiology. 1990 Oct;73(4):644-55. doi: 10.1097/00000542-199010000-00010. PMID 2221433
- [Background] Mangano DT. Perioperative cardiac morbidity. Anesthesiology. 1990 Jan;72(1):153-84. doi: 10.1097/00000542-199001000-00025. No abstract available. PMID 2404426
- [Background] Krupski WC, Layug EL, Reilly LM, Rapp JH, Mangano DT. Comparison of cardiac morbidity rates between aortic and infrainguinal operations: two-year follow-up. Study of Perioperative Ischemia Research Group. J Vasc Surg. 1993 Oct;18(4):609-15; discussion 615-7. PMID 8411468
- [Background] Knight AA, Hollenberg M, London MJ, Mangano DT. Myocardial ischemia in patients awaiting coronary artery bypass grafting. Am Heart J. 1989 Jun;117(6):1189-95. doi: 10.1016/0002-8703(89)90395-5. PMID 2786326
- [Background] Knight AA, Hollenberg M, London MJ, Tubau J, Verrier E, Browner W, Mangano DT. Perioperative myocardial ischemia: importance of the preoperative ischemic pattern. Anesthesiology. 1988 May;68(5):681-8. PMID 3259409
- [Background] O'Kelly BF, Tubau JF, Knight AA, London MJ, Verrier ED, Mangano DT. Measurement of left ventricular contractility using transesophageal echocardiography in patients undergoing coronary artery bypass grafting. The Study of Perioperative Ischemia (SPI) Research Group. Am Heart J. 1991 Oct;122(4 Pt 1):1041-9. doi: 10.1016/0002-8703(91)90470-3. PMID 1927855
- [Background] Leung JM. The role of hemodynamics in perioperative myocardial ischemia. Int Anesthesiol Clin. 1992 Winter;30(1):63-79. doi: 10.1097/00004311-199200000-00005. No abstract available. PMID 1577543
- [Background] Massie BM, Mangano DT. Assessment of perioperative risk: have we put the cart before the horse. J Am Coll Cardiol. 1993 May;21(6):1353-6. doi: 10.1016/0735-1097(93)90308-n. No abstract available. PMID 8473641
- [Background] Hollenberg M, Mangano DT. Therapeutic approaches to postoperative ischemia. The Study of Perioperative Ischemia Research Group. Am J Cardiol. 1994 Mar 10;73(6):30B-33B. doi: 10.1016/0002-9149(94)90263-1. PMID 8141077
- [Background] Mangano DT, Layug EL, Wallace A, Tateo I. Effect of atenolol on mortality and cardiovascular morbidity after noncardiac surgery. Multicenter Study of Perioperative Ischemia Research Group. N Engl J Med. 1996 Dec 5;335(23):1713-20. doi: 10.1056/NEJM199612053352301. PMID 8929262
- [Background] Halm EA, Browner WS, Tubau JF, Tateo IM, Mangano DT. Echocardiography for assessing cardiac risk in patients having noncardiac surgery. Study of Perioperative Ischemia Research Group. Ann Intern Med. 1996 Sep 15;125(6):433-41. doi: 10.7326/0003-4819-125-6-199609150-00001. PMID 8779454